CLINICAL TRIAL: NCT01665183
Title: Phase 1 Trial of ADI-PEG 20 Plus Cisplatin in Patients With Metastatic Melanoma or Other Advanced Solid Malignancies
Brief Title: Ph 1 Trial of ADI-PEG 20 Plus Cisplatin in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLARIS2012-005
Record Dates: First submitted 2012-08-08; First posted 2012-08-15 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Cutaneous Melanoma, Uveal Melanoma, Ovarian Carcinoma or Other Advanced Solid Tumors
Keywords: argininosuccinate synthetase; arginine; arginine deiminase
MeSH Terms: conditions — Melanoma; Uveal Melanoma; Ovarian Neoplasms | interventions — ADI PEG20; Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADI-PEG 20 (Experimental): arginine deiminase formulated with polyethylene glycol
  Interventions: Drug: ADI-PEG 20

INTERVENTIONS:
Drug: ADI-PEG 20
  Other Names: arginine deiminase formulated with polyethylene glycol

SUMMARY:
Certain cancers require the amino acid arginine. Arginine deiminase (ADI) is an enzyme from microbes that degrades arginine. ADI has been formulated with polyethylene glycol, and has been used to treat patients that have cancers that require arginine. In this study, ADI will be combined with the well known chemotherapy cisplatin, and the safety and potential efficacy of this combination will be explored in patients with cancers that require arginine.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of advanced solid tumor (dose escalation component) or metastatic melanoma (uveal or cutaneous) (doses escalation and MTD expansion components) or platinum-resistant (tumor progression within a year after the completion of platinum-based therapy) ovarian carcinoma (high grade serous, endometrial or poorly differentiated endometrioid) or HCC that has failed treatment with sorafenib or did not tolerate sorafenib or refused sorafenib, or HCC with coexistent BCT that has or has not been treated with chemotherapy, or BCT that has or has not been treated with chemotherapy. For HCC and HCC with coexistent BCT, cirrhotic status of Child-Pugh grade A-B7 must be present. Child-Pugh status should be determined based on clinical findings and laboratory data during the screening period (Appendix C). Subjects on anti-coagulants are to receive 1 point for their INR status, as they are presumed to have a <1.7 baseline PT/INR.
2. Ovarian cancer, or HCC, or HCC with coexistent BCT, or BCT only tissue either from an archived specimen or from a new biopsy of sufficient amount and quality should be available for IHC determination of ASS status to be performed retrospectively for the ovarian cancer, or HCC, or HCC with coexistent BCT, or BCT only cohorts. Subjects with no tissue available would require a biopsy.
3. Unresectable disease or patient refused surgery.
4. Progressive disease if treated with chemotherapy, radiotherapy, surgery or immunotherapy. If prior radiation was given, the measurable disease should be outside the radiation port. Unequivocal progression of HCC/BTC lesions previously treated with catheter-based therapy including transarterial chemoembolization or radioembolization is allowed.
5. Measurable disease as assessed by RECIST 1.1 criteria (Appendix A).
6. Age ≥ 18 years.
7. ECOG performance status of 0 - 1.
8. No prior systemic therapy, immunotherapy, investigational agent, chemoembolization, radioembolization or radiation therapy within the last 4 weeks.
9. Fully recovered from any prior surgery and no major surgery within 4 weeks of initiating treatment, except for gamma knife which can take place within 2 weeks. Surgery for placement of vascular access devices is acceptable.

Exclusion Criteria:

1. Serious infection requiring treatment with systemically administered antibiotics at the time of study entrance, or an infection requiring systemic antibiotic therapy within 7 days prior to the first dose of study treatment. For the HCC, HCC/BTC and BTC subgroups hepatitis C infection and hepatitis B infection if controlled with antiviral therapy are allowable.
2. Pregnancy or lactation.
3. Expected non-compliance.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV), cardiac arrhythmia, or psychiatric illness, social situations that would limit compliance with study requirements.
5. Subjects who have had any anticancer treatment prior to entering the study and have not recovered to baseline (except alopecia) or ≤ Grade 1 AEs, or deemed irreversible from the effects of prior cancer therapy. AEs > Grade 1 that are not considered a safety risk by the Sponsor and investigator may be allowed upon agreement with both.
6. Subjects with history of another primary cancer, including co-existent second malignancy, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor with no known active disease present in the opinion of the investigator will not affect patient outcome in the setting of current cancer diagnosis.
7. Subjects who had been treated with ADI-PEG 20 previously.
8. History of seizure disorder not related to underlying cancer.
9. Known HIV positivity (testing not required).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events. | Course of study.

SECONDARY OUTCOMES:
Number of participants with objective responses. | Course of study.

CONTACTS AND LOCATIONS:
Overall Officials: Siqing Fu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- MD Anderson Cancer Center, Houston, Texas, United States
- NCKUH, Tainan, Taiwan